CLINICAL TRIAL: NCT03187756
Title: Phase II Study of Nonmyeloablative Peripheral Blood Stem Cell Transplant With High-dose Posttransplantation Cyclophosphamide in Hematopoietic Malignancies Including Those That Are Challenging to Engraft
Brief Title: Study of Nonmyeloablative Peripheral Blood Stem Cell Transplant With High-dose Posttransplantation Cyclophosphamide in Hematopoietic Malignancies Including Those That Are Challenging to Engraft
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Procedure has become standard of care - protocol is no longer necessary
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00042
Record Dates: First submitted 2017-06-02; First posted 2017-06-15 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Hematopoietic Malignancies
Keywords: Hematopoietic Malignancies; Nonmyeloablative Peripheral Blood Stem Cell Transplant; Posttransplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cyclophosphamide (Experimental)
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Shortened duration immunosuppression following nonmyeloablative peripheral blood stem cell transplant with high dose post transplantation cyclophosphamide in malignancies to engraft.

SUMMARY:
This is an open label phase II single arm study of peripheral blood stem cell transplantation and posttransplantation cyclophosphamide, using HLA full match or haploidentical related donors, in hematological malignancies including those difficult to engraft. The objective of this study is to evaluate the safety and feasibility in nonmyeloablative, partially HLA-mismatched or HLA-matched PBSC transplant from haploidentical donors or fully matched donors with post-grafting immunosuppression that includes high-dose cyclophosphamide, tacrolimus, and Mycophenolate mofetil (MMF).

DETAILED DESCRIPTION:
Primary Objective Estimate event free survival (EFS) (relapse, progression, or death) rate one year after transplant.

Secondary Objectives:

1. Estimate the cumulative incidences of severe acute grade III or higher GVHD, chronic GVHD (overall and by extent)
2. Estimate the cumulative incidence of systemic steroid initiation,
3. Summarize the graft failure frequency,
4. Summarize the kinetics of neutrophil and platelet recovery, and kinetics of donor chimerism in unsorted and CD3+ sorted peripheral blood.
5. Summarize major toxicities and complications associated with the transplantation procedure selected toxicities.

Exploratory Objectives:

Explore the association between the amount of donor T cell chimerism at ~ Day 28 and patient/graft characteristics (e.g., prior therapies, graft cell dose) and transplantation outcomes (sustained engraftment, relapse or progression, GVHD).

ELIGIBILITY:
Inclusion Criteria:

The following are eligibility for study entry and transplantation.

* Presence of a suitable related, HLA-haploidentical or HLA-matched stem cell donor
* The donor and recipient must be identical at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. A minimum match of 5/10 is therefore required for related donors, and will be considered sufficient evidence that the donor and recipient share one HLA haplotype.
* Eligible diagnoses:
* Myelodysplastic syndrome (MDS) including chronic myelomonocytic leukemia [CMML] with at least one poor risk factor
* No active extramedullary leukemia or known active CNS involvement by malignancy. Such disease treated into remission is permitted.
* Any previous autologous HSCT must have occurred at least 3 months prior to start of conditioning
* No previous allogeneic HSCT
* Adequate end-organ function Note: Infection is permitted if there is evidence of response to medication. Eligibility of HIV infected patients will be determined on a case-by-case basis.
* ECOG performance status < 2 or Karnofsky or Lansky score > 60.
* Age > 18 years and older.
* Not pregnant or breast-feeding.
* No uncontrolled infection.

Eligible diagnoses:

* Myelodysplastic syndrome (MDS) including chronic myelomonocytic leukemia [CMML] with at least one of the following poor-risk features
* SLL or CLL with 17p deletion, or with progression < 6 months after second or greater treatment regimen. Must have the following to be an acceptable candidate as well:

  * < 20% of bone marrow cellularity involved by SLL/CLL (to lower risk of graft rejection)
  * No lymph nodes > 5 cm in any dimension
  * No massive splenomegaly, defined as > 6 cm below the left costal margin
* T-cell PLL in PR or better prior to transplantation. Must also have < 20% of bone marrow cellularity involved by PLL (to lower risk of graft rejection).
* Interferon- or tyrosine kinase-refractory CML in first chronic phase, TKI-intolerant CML in first chronic phase, or CML in second or subsequent chronic phase
* Philadelphia chromosome negative myeloproliferative disease (including myelofibrosis)

  o Intermediate-2 or High risk score by DIPSS Plus is required for a diagnosis of myelofibrosis
* Multiple myeloma or plasma cell leukemia with a PR or better to the last treatment regimen, based on the International Myeloma Working Group (IMWG) criteria.49
* Hematologic malignancy in complete remission with minimal residual disease (MRD) non detectable OR detectable by conventional cytogenetics, FISH, flow cytometry, or molecular testing or hematologic malignancies in partial remission

Donor eligibility

* Donors must be either:
* HLA-haploidentical or HLA-identical relatives of the patient based on allele or allele group level typing as defined in Section 4.1.
* Medically fit to and willing to donate
* Lack of recipient anti-donor HLA antibody
* Has not donated blood products to patient

Exclusion Criteria:

* Any individual that does not meet the eligibility criteria for transplantation or donor eligibility will not be a part of this trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer Al-Homsi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide: Cy 50 mg/kg IV, over approximately 1-2 hours (depending on volume), is given on Day 3 posttransplantation (ideally between 60 and 72 hours after marrow infusion) and on Day 4 (approximately 24 hours after Day 3 Cy).
Period: Overall Study
Arm/Group | Cyclophosphamide
Started | 6
Completed | 2
Not Completed | 4
Not completed — Termination of study | 4

BASELINE CHARACTERISTICS:
Population: 6 participants enrolled, but only 2 participants completed
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: Years] | 51 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS)
Description: Estimate the one year after transplantation event free survival (EFS) rate using a Kaplan-Meier curve with a 90% confidence interval. An event for EFS is defined as the first of any of the following failures: relapse or disease progression or death from any cause
Time Frame: One Year
Population: 2 participants reached the 1 year time point but disease assessment was completed for only 1 subject (complete remission).
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Participants With Chronic GVHD and Grades I-IV GVHD
Description: Acute GVHD is graded by standard criteria, and all suspected cases of acute GVHD will be confirmed histologically by biopsy of an affected organ. The severity of acute GVHD is determined by an assessment of the degree of involvement of the skin, liver, and gastrointestinal tract. Grade I is characterized as mild disease (skin involvement alone), Grade II as moderate, Grade III as severe (involvement of any organ system), and Grade IV as life-threatening. The diagnosis of a chronic GVHD per NIH criteria requires a) at least 1 diagnostic manifestation or b) 1 distinctive manifestation confirmed by biopsy or testing of the same or other involved organ.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 6
Participants
  chronic GVHD | 0
  acute grade IV GVHD | 0
  acute grade III GVHD | 0
  acute grade II GVHD | 0
  acute grade I GVHD | 2

3. Secondary Outcome: Number of Major Toxicities and Complications Associated With Transplantation Procedure
Description: Summarize major toxicities and complications associated with the transplantation procedure
Time Frame: 1 year
Population: While AE data was reported (see AE / SAE section), due to termination of the study, relationship of major AEs to transplant procedures was unable to be assessed. Therefore, this information cannot be reported.
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 0

4. Secondary Outcome: Cumulative Incidences of Systemic Steroid Initiation
Description: Estimate the cumulative incidence of systemic steroid initiation, by 1 year after HSCT. This is will be reported as number of participants who started steroids over the course of the study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 6
Participants | 6

5. Secondary Outcome: Graft Failure Frequency
Description: Graft failure and death, or graft failure, death and treatment of relapse/progressions. This will be reported as the number of participants with graft failures.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 6
Participants | 0

6. Secondary Outcome: Time to Neutrophil Recovery
Description: Neutrophil recovery is defined as post-nadir ANC greater than or equal to 500/mm3 for three consecutive measurements on different days. The first of the three days will be designated as the day of neutrophil recovery.
Time Frame: 1 year
Measure: Mean (Full Range); unit: days
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 6
days | 24.17 [17 to 31]

7. Secondary Outcome: Time to Platelet Recovery
Description: Platelet recovery is defined as sustained platelet count greater than or equal to 20,000/mm3 or greater than or equal to 50,000/mm3 with no platelet transfusions in the preceding seven days. The first of three consecutive measurements on different days will be designated as the day of initial platelet recovery.
Time Frame: 1 year
Measure: Mean (Full Range); unit: days
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 6
days | 9.4 [1 to 24]

ADVERSE EVENTS:
Time Frame: The time frame for adverse event data collection was 13 months.
Description: All adverse events occurring during the study period were reported. The clinical course of each event was followed up until resolution, stabilization, or until it was determined that the study treatment or participation was not the cause.
Arm/Group | Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide (N=6)
Cytomegalovirus (Infections and infestations) | 1 (1)
Fever (General disorders) | 4 (5)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide (N=6)
Adenovirus (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Vomiting (Metabolism and nutrition disorders) | 1 (1)
Uticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Upper Respiratory Tract Infection (URI) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper GI Stage 1 Acute GVHD (Gastrointestinal disorders) | 1 (1)
Transaminitis MILD (Hepatobiliary disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
superficial thrombophlebitis (Left Arm) (Blood and lymphatic system disorders) | 1 (1)
Sore Throat (General disorders) | 1 (1)
Skin Stage 1 Acute GVHD (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinovirus (Infections and infestations) | 1 (1)
Rectal Mucositis (Gastrointestinal disorders) | 1 (1)
Radiation Enteritis (Gastrointestinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Parainfluenza (Infections and infestations) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Palmar Plantar Erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Norovirus (Infections and infestations) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Neoropathy (Nervous system disorders) | 1 (1)
Neck Pain (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nasal Congestion (General disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Intermittent Tremor (General disorders) | 1 (1)
Intermittent Increased Serum Creatinine (Hepatobiliary disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 4 (4)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Headache (General disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03187756/Prot_SAP_000.pdf